CLINICAL TRIAL: NCT06025123
Title: Prehospital Resuscitation Intranasal Cooling Effectiveness Survival Study 2 (PRINCESS2)
Brief Title: Prehospital Resuscitation Intranasal Cooling Effectiveness Survival Study 2
Acronym: PRINCESS2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Per Nordberg, Senior consultant in cardiology and intensive care, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-02446-01
Record Dates: First submitted 2023-02-01; First posted 2023-09-06 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Hypothermia; Ventricular Fibrillation
Keywords: Therapeutic hypothermia; transnasal cooling; neurologic outcome; ultrafast hypothermia; prehospital; ECPR
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Hypothermia; Ventricular Fibrillation

STUDY DESIGN:
Intervention Model Description: Patients will be randomized by EMS personnel at the scene of cardiac arrest to either a) intervention: early transnasal evaporative cooling initiated within 20 minutes from EMS arrival, and subsequent systemic hypothermia at 33°C for 24 h and fever control for 72 h in the ICU, or b) control: standard ACLS (advanced cardiac life support) and fever control (normothermia) for 72 h in the ICU.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Patients in the intervention group will be treated with hypothermia, which makes blinding for care provider and next of kin difficult in the intervention phase (first 36 h). Participants will be informed of which group the were assigned to if they regained consciousness. The study personnel assessing neurologic outcome at discharge and at 90 days will be blinded for which study group the participant belongs to. In addition, the physician performing the prognostication at 72 hours from cardiac arrest will be a neurologist, intensivist or other specialist experienced and will be blinded for group allocation, but not for relevant clinical data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early transnasal evaporative cooling with the RhinoChill device (Experimental): Early transnasal evaporative cooling initiated during ACLS at the scene of the cardiac arrest within 20 minutes from EMS arrival and subsequent hypothermia at 33ºC for 24 hours and fever control for 72 hours at the ICU
  Interventions: Device: Early transnasal evaporative cooling with the RhinoChill device
- Standard of care (No Intervention): Standard advanced cardiac life support, subsequent fever control (Normothermia) for 72 hours at ICU

INTERVENTIONS:
Device: Early transnasal evaporative cooling with the RhinoChill device — Early prehospital transnasal evaporative cooling followed by systemic hypothermia to 33 degrees Celsius for 24 hours and fever control for 72 hours
  Arms: Early transnasal evaporative cooling with the RhinoChill device

SUMMARY:
The aim of this clinical trial is to study the impact of ultra-early transnasal evaporative cooling after cardiac arrest and subsequent hypothermia at hospital, on survival with complete neurologic recovery, compared to currently recommended normothermia. The study population will consist of patients 18-79 years old, with out-of-hospital cardiac arrest with initial shockable rhythm.

The main research question it aims to answer is whether there is a difference in survival with complete neurologic recovery at 90 days after cardiac arrest between the group of patients that received ultra-early cooling, compared to the group that was treated with normothermia.

Participants will be randomized to two groups. One group (the intervention group) will receive ultra-early trans-nasal evaporative cooling initiated by EMS personnel at the scene of the cardiac arrest, and subsequent systemic hypothermia for 24 hours at hospital arrival. The other group (the control group), will receive standard of care (advanced cardiac life support and normal body temperature (normothermia)).

ELIGIBILITY:
INCLUSION CRITERIA:

Patients ≥18 years that meet all of the following inclusion criteria:

1. Adult out-of-hospital cardiac arrest patients with initial shockable rhythm
2. Unconsciousness defined as Glasgow Coma Scale < 8
3. Inclusion within 20 minutes from EMS arrival

EXCLUSION CRITERIA:

Patients are not eligible if they meet one or more of the following criteria:

1. Age ≥ 80 years
2. Obvious non-cardiac causes to cardiac arrest
3. Obvious already hypothermic
4. Obvious barrier to placing intra nasal catheters
5. Have a known Do Not Attempt to Resuscitate (DNAR) order or other limitations in care
6. Have a known terminal disease
7. Known or clinically apparent pregnancy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1022 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients surviving with complete neurologic recovery at 90 days defined as modified Rankin scale (mRs) of 0-1. | Day 90
  The modified Rankin Scale is a scoring system on neurologic function ranging from 0-6, where 0 means no symtoms at all, higher numbers indicating increasing neurologic disabilities and 6 equals death.

SECONDARY OUTCOMES:
Proportion of patients with sustained ROSC (return of spontaneous circulation) and admitted alive to hospital | Day 1
Proportion of patients alive at hospital discharge | Day 1-90
Proportion of patients with Modified Rankin scale 0-3 at hospital discharge | Day 1-90
  The modified Rankin Scale is a scoring system on neurologic function ranging from 0-6, where 0 means no symtoms at all, higher numbers indicating increasing neurologic disabilities and 6 equals death.
Proportion of patients alive at 90 days | Day 90
Proportion of patients with Modified Rankin scale 0-3 at 90 days | Day 90
  The modified Rankin Scale is a scoring system on neurologic function ranging from 0-6, where 0 means no symtoms at all, higher numbers indicating increasing neurologic disabilities and 6 equals death.
Device related adverse event rate within the first 24 hours | Day 1
  Safety
Composite serious adverse event rate within the first 7 days | Day 1-7
  Safety
Proportion of patients with new cardiac arrest prior to hospital admission | Day 1
  Safety

OTHER OUTCOMES:
Hospital-free days alive at 90 days | Day 90
Distribution of modified Rankin scale at 90 days | Day 90
  The modified Rankin Scale is a scoring system on neurologic function ranging from 0-6, where 0 means no symtoms at all, higher numbers indicating increasing neurologic disabilities and 6 equals death.
Distribution of Cerebral Performance Category scale at 90 days | Day 90
  The Cerebral Performance Category (CPC) scale is a measure for neurologic function. It ranges from 1-5, where 1 equals no or minimal neurologic disabilities, and 5 equals death.
Proportion of patients alive after 1 year | Day 365
Proportion of patients with Modified Rankin scale 0-1 at 1 year | Day 365
  The modified Rankin Scale is a scoring system on neurologic function ranging from 0-6, where 0 means no symtoms at all, higher numbers indicating increasing neurologic disabilities and 6 equals death.
Quality of life assessed with EQ-5D-5L at 90 days | Day 90
  EQ-5D is a a measure of health status and quality of life defined in terms of mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is divided into three levels; no problems, some or moderate problems or extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Per Nordberg, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (11):
- University Hospital Vienna, Vienna, Austria
- Belgium (3):
  - CHU Saint-Pierre, Brussels
  - Erasme University Hospital, Brussels
  - Europe Hospitals St Elizabeth, Brussels
- University Hospital Freiburg, Freiburg im Breisgau, Germany
- Department of Anesthesiology, Intensive Care and Emergency, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy
- Ljubljana University Medical Centre, Ljubljana, Slovenia
- Spain (2):
  - Hospital Universitario La Paz, Madrid
  - San Carlos Clinical Hospital, Madrid
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Södersjukhuset, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dillenbeck E, Hollenberg J, Holzer M, Busch HJ, Nichol G, Radsel P, Belohlavec J, Torres EC, Lopez-de-Sa E, Rosell F, Ristagno G, Forsberg S, Annoni F, Svensson L, Jonsson M, Backstrom D, Gellerfors M, Awad A, Taccone FS, Nordberg P. The design of the PRINCESS 2 trial: A randomized trial to study the impact of ultrafast hypothermia on complete neurologic recovery after out-of-hospital cardiac arrest with initial shockable rhythm. Am Heart J. 2024 May;271:97-108. doi: 10.1016/j.ahj.2024.02.020. Epub 2024 Feb 28. PMID 38417773

DOCUMENTS (2):
  • Study Protocol (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT06025123/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT06025123/SAP_001.pdf